CLINICAL TRIAL: NCT03335527
Title: Impact of Low-Dose Dexmedetomidine on Sleep Quality in Mechanical Ventilation Patients After Surgery in Intensive Care Unit: a Pilot Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Impacts of Low-Dose Dexmedetomidine on Sleep Quality in Mechanically Ventilated ICU Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2017[13]
Record Dates: First submitted 2017-11-02; First posted 2017-11-07 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Aged; Postoperative Period; Intensive Care Units; Mechanical Ventilation Complication; Sleep Disorders; Dexmedetomidine
Keywords: Aged; Postoperative period; Intensive Care Unit; Mechanical ventilation; Sleep quality; Dexmedetomidine
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Experimental): Dexmedetomidine is infused at a rate of 0.1 ug/kg/h during mechanical ventilation, for a maximum of 3 days
  Interventions: Drug: Dexmedetomidine
- Placebo group (Placebo Comparator): Placebo (normal saline) is infused at a same rate as in the dexmedetomidine group during mechanical ventilation, for a maximum of 3 days
  Interventions: Drug: Placebo (normal saline)

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine is administered as a continuous intravenous infusion at a rate of 0.1-0.2 ug/kg/h (0.025-0.05 ml/kg/h) from study recruitment in the ICU during mechanical ventilation, for no more than 72 hours.
  Other Names: Dexmedetomidine hydrochloride
  Arms: Dexmedetomidine group
Drug: Placebo (normal saline) — Placebo (normal saline) is administered as a continuous intravenous infusion at a rate of 0.025-0.05 ml/kg/h from study recruitment in the ICU during mechanical ventilation, for no more than 72 hours.
  Other Names: Normal saline
  Arms: Placebo group

SUMMARY:
Sleep disturbances frequently occur in intensive care unit (ICU) patients undergoing mechanical ventilation. In a previous study, sedative dose dexmedetomidine (median 0.6 microgram/kg/h) improved sleep quality in mechanically ventilated patients. However, for mechanically ventilated patients, light sedation is better than deep sedation for the outcomes, which is manifested as shortened length of ICU stay, shortened duration of mechanical ventilation, and decreased mortality. In a recent study of the investigators, non-sedative low-dose dexmedetomidine (0.1 microgram/kg/h) improved sleep quality in non-mechanically ventilated elderly patients admitted to the ICU after surgery. The investigators hypothesize that, in mechanically ventilated patients who are admitted to the ICU after surgery, low-dose dexmedetomidine may also improve sleep quality.

DETAILED DESCRIPTION:
Sleep is severely disturbed in mechanically ventilated ICU patients, especially those after surgery. Polysomnographic studies performed in these patients demonstrated a severe increase in sleep fragmentation, prolonged N1 and N2 sleep, reduced N3 and REM sleep, and an abnormal distribution of sleep because almost half of the total sleep time occurred during the daytime. Patients reported little or no sleep, poor sleep quality, frequent awakening, and daytime sleep.

Many factors are responsible for sleep disturbance in postoperative ICU patients with mechanical ventilation, these include the severity of surgical stress and illness, ICU environment, mechanical ventilation, pain, sedatives and analgesics, and various other therapy. Sleep disturbances produce harmful effects on postoperative outcomes. It is associated with increased prevalence of delirium, cardiac events and worse functional recovery. Moreover, patients with sleep disturbances are more sensitive to pain.

Unlike other sedative agents, dexmedetomidine exerts its sedative effects through an endogenous sleep-promoting pathway and produces a N2 sleep-like state. In mechanically ventilated ICU patients, nighttime infusion of sedative dose of dexmedetomidine (median 0.6 microgram/kg/h) preserved the day-night cycle of sleep and improved the sleep architecture by increasing sleep efficiency and stage N2 sleep.

Studies showed that, in mechanically ventilated patients, light sedation is better than deep sedation for patients' outcomes, including shortened duration of ventilation and length of ICU stay, and decreased mortality. Some studies even showed that no sedation (analgesia only) is better than sedation. In a recent study of non mechanical ventilated elderly patients who were admitted to the ICU after surgery, non-sedative low-dose dexmedetomidine infusion (at a rate of 0.1 microgram/kg/h during the night on the day of surgery) increased the percentage of stage N2 sleep (and decreased the percentage of N1 sleep), prolonged the total sleep time, increased the sleep efficiency, and improved the subjective sleep quality.

The investigators hypothesize that, in mechanically ventilated patients who were admitted to the ICU after surgery, low-dose dexmedetomidine infusion may also improve sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older;
* admitted to the ICU after surgery;
* with an expected duration of mechanical ventilation of more than 12 hours (admitted before 21:00 on the day of surgery and extubated after 06:00 on the first day after surgery).

Exclusion Criteria:

* refused to participate;
* aged less than 18 years;
* pregnant;
* preoperative history of schizophrenia, epilepsy, parkinsonism, or myasthenia gravis;
* inability to communicate in the preoperative period (coma, profound dementia, or language barrier);
* brain injury or neurosurgery;
* known preoperative left ventricular ejection fraction less than 30%, sick sinus syndrome, severe sinus bradycardia (<50 beats per min), or second degree or greater atrioventricular block without pacemaker, systolic blood pressure less than 90 mmHg despite continuous infusions of vasopressors before the start of study drugs infusion;
* serious hepatic dysfunction (Child-Pugh class C);
* serious renal dysfunction (undergoing dialysis before surgery);
* less likelihood to survive for more than 24 hours;
* preoperative history of sleep disorders (requirement of hypnotics/sedatives during the last month) or history of obstructive sleep apnea syndrome (diagnosed with obstructive sleep apnea);
* allergy to the study drugs;
* other conditions that are considered unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Sleep quality during the night of surgery. | Assessed at 08:00 on the first day after surgery.
  Sleep quality assessed with Richards-Campbell Sleep Questionnaire at 08:00 on the first day after surgery.

SECONDARY OUTCOMES:
Incidence of delirium within the first 7 days after surgery. | Assessed twice daily during the first 7 days after surgery.
  Assessment twice daily (in the morning from 06:00 to 10:00 and in the evening from 18:00 to 20:00) with the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU).
Sleep quality within the first 7 days after surgery. | Assessed once daily during the first 7 days after surgery.
  Assessment once daily (at 08:00) with Richards-Campbell Sleep Questionnaire (RCSQ).
Total sleep time | Monitored with polysomnograph during the night of surgery.
  Total sleep time
Sleep efficiency | Monitored with polysomnograph during the night of surgery.
  Sleep efficiency
Fragmented sleep index | Monitored with polysomnograph during the night of surgery.
  Fragmented sleep index
Percentages of sleep stages | Monitored with polysomnograph during the night of surgery.
  Percentages of stage 1 non-rapid sleep movement sleep (N1), N2, N3 and rapid eye movement (REM) sleep.
Duration of mechanical ventilation. | From ICU admission to 30 days after surgery.
  Duration of mechanical ventilation.
Length of stay in the ICU. | From ICU admission to 30 days after surgery.
  Length of stay in the ICU.
Length of stay in the hospital after surgery. | From date of surgery to 30 days after surgery.
  Length of stay in the hospital after surgery.
Occurrence of postoperative complications. | From date of surgery to 30 days after surgery.
  Occurrence of complications other than delirium within 30 days after surgery.
All-cause 30-day mortality. | On the 30th day after surgery.
  All-cause 30-day mortality.
30-day cognitive function. | On the 30th day after surgery.
  Assessment with Telephone Interview for Cognitive Status-modified (TICS-m) in 30-day survivors.
30-day quality of life. | On the 30th day after surgery.
  Assessment with WhoQOL-Bref.
30-day sleep quality. | On the 30th day after surgery.
  Assessment with Pittsburgh Sleep Quality Index (PSQI).

OTHER OUTCOMES:
Pain intensity. | Assessed during the first 7 days after surgery.
  Assessment twice daily (in the morning from 06:00 to 10:00 and in the evening from 18:00 to 20:00) with the Numeric Rating Scale (NRS, an 11 point scale where 0 indicated no pain and 10 indicated the worst possible pain) at movement or the Behavior Pain Scale (BPS, an 12 point scale where 3 indicated no pain and 12 indicated the worst possible pain) at rest.
Score of Acute Physiology and Chronic Health Evaluation II (APACHE II). | Assessed within 24 hours after ICU admission.
  Score of Acute Physiology and Chronic Health Evaluation II (APACHE II).
Percentage of time within the target of sedation during mechanical ventilation. | During mechanical ventilation, for a maximum of 3 days.
  Percentage of time within the target of sedation (Richmond Agitation-Sedation Scale -1~-2) during mechanical ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Friese RS. Sleep and recovery from critical illness and injury: a review of theory, current practice, and future directions. Crit Care Med. 2008 Mar;36(3):697-705. doi: 10.1097/CCM.0B013E3181643F29. PMID 18176314
- [Background] Elliott R, McKinley S, Cistulli P. The quality and duration of sleep in the intensive care setting: an integrative review. Int J Nurs Stud. 2011 Mar;48(3):384-400. doi: 10.1016/j.ijnurstu.2010.11.006. Epub 2010 Dec 24. PMID 21185560
- [Background] Cooper AB, Thornley KS, Young GB, Slutsky AS, Stewart TE, Hanly PJ. Sleep in critically ill patients requiring mechanical ventilation. Chest. 2000 Mar;117(3):809-18. doi: 10.1378/chest.117.3.809. PMID 10713011
- [Background] Parsons EC, Kross EK, Caldwell ES, Kapur VK, McCurry SM, Vitiello MV, Hough CL. Post-discharge insomnia symptoms are associated with quality of life impairment among survivors of acute lung injury. Sleep Med. 2012 Sep;13(8):1106-9. doi: 10.1016/j.sleep.2012.05.010. Epub 2012 Jul 2. PMID 22763017
- [Background] Combes A, Costa MA, Trouillet JL, Baudot J, Mokhtari M, Gibert C, Chastre J. Morbidity, mortality, and quality-of-life outcomes of patients requiring >or=14 days of mechanical ventilation. Crit Care Med. 2003 May;31(5):1373-81. doi: 10.1097/01.CCM.0000065188.87029.C3. PMID 12771605
- [Background] Granja C, Lopes A, Moreira S, Dias C, Costa-Pereira A, Carneiro A; JMIP Study Group. Patients' recollections of experiences in the intensive care unit may affect their quality of life. Crit Care. 2005 Apr;9(2):R96-109. doi: 10.1186/cc3026. Epub 2005 Jan 31. PMID 15774056
- [Background] Aurell J, Elmqvist D. Sleep in the surgical intensive care unit: continuous polygraphic recording of sleep in nine patients receiving postoperative care. Br Med J (Clin Res Ed). 1985 Apr 6;290(6474):1029-32. doi: 10.1136/bmj.290.6474.1029. PMID 3921096
- [Background] Friese RS, Diaz-Arrastia R, McBride D, Frankel H, Gentilello LM. Quantity and quality of sleep in the surgical intensive care unit: are our patients sleeping? J Trauma. 2007 Dec;63(6):1210-4. doi: 10.1097/TA.0b013e31815b83d7. PMID 18212640
- [Background] Gehlbach BK, Chapotot F, Leproult R, Whitmore H, Poston J, Pohlman M, Miller A, Pohlman AS, Nedeltcheva A, Jacobsen JH, Hall JB, Van Cauter E. Temporal disorganization of circadian rhythmicity and sleep-wake regulation in mechanically ventilated patients receiving continuous intravenous sedation. Sleep. 2012 Aug 1;35(8):1105-14. doi: 10.5665/sleep.1998. PMID 22851806
- [Background] Elliott R, McKinley S, Cistulli P, Fien M. Characterisation of sleep in intensive care using 24-hour polysomnography: an observational study. Crit Care. 2013 Mar 18;17(2):R46. doi: 10.1186/cc12565. PMID 23506782
- [Background] Slatore CG, Goy ER, O'hearn DJ, Boudreau EA, O'Malley JP, Peters D, Ganzini L. Sleep quality and its association with delirium among veterans enrolled in hospice. Am J Geriatr Psychiatry. 2012 Apr;20(4):317-26. doi: 10.1097/JGP.0b013e3182487680. PMID 22367162
- [Background] Kjolhede P, Langstrom P, Nilsson P, Wodlin NB, Nilsson L. The impact of quality of sleep on recovery from fast-track abdominal hysterectomy. J Clin Sleep Med. 2012 Aug 15;8(4):395-402. doi: 10.5664/jcsm.2032. PMID 22893770
- [Background] Fernandes NM, Nield LE, Popel N, Cantor WJ, Plante S, Goldman L, Prabhakar M, Manlhiot C, McCrindle BW, Miner SE. Symptoms of disturbed sleep predict major adverse cardiac events after percutaneous coronary intervention. Can J Cardiol. 2014 Jan;30(1):118-24. doi: 10.1016/j.cjca.2013.07.009. Epub 2013 Oct 16. PMID 24140074
- [Background] Finan PH, Goodin BR, Smith MT. The association of sleep and pain: an update and a path forward. J Pain. 2013 Dec;14(12):1539-52. doi: 10.1016/j.jpain.2013.08.007. PMID 24290442
- [Background] Kanji S, Mera A, Hutton B, Burry L, Rosenberg E, MacDonald E, Luks V. Pharmacological interventions to improve sleep in hospitalised adults: a systematic review. BMJ Open. 2016 Jul 29;6(7):e012108. doi: 10.1136/bmjopen-2016-012108. PMID 27473952
- [Background] Stanchina ML, Abu-Hijleh M, Chaudhry BK, Carlisle CC, Millman RP. The influence of white noise on sleep in subjects exposed to ICU noise. Sleep Med. 2005 Sep;6(5):423-8. doi: 10.1016/j.sleep.2004.12.004. Epub 2005 Mar 31. PMID 16139772
- [Background] Freedman NS, Gazendam J, Levan L, Pack AI, Schwab RJ. Abnormal sleep/wake cycles and the effect of environmental noise on sleep disruption in the intensive care unit. Am J Respir Crit Care Med. 2001 Feb;163(2):451-7. doi: 10.1164/ajrccm.163.2.9912128. PMID 11179121
- [Background] Parthasarathy S, Tobin MJ. Effect of ventilator mode on sleep quality in critically ill patients. Am J Respir Crit Care Med. 2002 Dec 1;166(11):1423-9. doi: 10.1164/rccm.200209-999OC. Epub 2002 Sep 5. PMID 12406837
- [Background] Fanfulla F, Ceriana P, D'Artavilla Lupo N, Trentin R, Frigerio F, Nava S. Sleep disturbances in patients admitted to a step-down unit after ICU discharge: the role of mechanical ventilation. Sleep. 2011 Mar 1;34(3):355-62. doi: 10.1093/sleep/34.3.355. PMID 21358853
- [Background] Trompeo AC, Vidi Y, Locane MD, Braghiroli A, Mascia L, Bosma K, Ranieri VM. Sleep disturbances in the critically ill patients: role of delirium and sedative agents. Minerva Anestesiol. 2011 Jun;77(6):604-12. PMID 21617624
- [Background] Weinhouse GL, Watson PL. Sedation and sleep disturbances in the ICU. Crit Care Clin. 2009 Jul;25(3):539-49, ix. doi: 10.1016/j.ccc.2009.04.003. PMID 19576529
- [Background] Gabor JY, Cooper AB, Crombach SA, Lee B, Kadikar N, Bettger HE, Hanly PJ. Contribution of the intensive care unit environment to sleep disruption in mechanically ventilated patients and healthy subjects. Am J Respir Crit Care Med. 2003 Mar 1;167(5):708-15. doi: 10.1164/rccm.2201090. PMID 12598213
- [Background] Schiza SE, Simantirakis E, Bouloukaki I, Mermigkis C, Arfanakis D, Chrysostomakis S, Chlouverakis G, Kallergis EM, Vardas P, Siafakas NM. Sleep patterns in patients with acute coronary syndromes. Sleep Med. 2010 Feb;11(2):149-53. doi: 10.1016/j.sleep.2009.07.016. Epub 2010 Jan 18. PMID 20083431
- [Background] Nelson LE, Lu J, Guo T, Saper CB, Franks NP, Maze M. The alpha2-adrenoceptor agonist dexmedetomidine converges on an endogenous sleep-promoting pathway to exert its sedative effects. Anesthesiology. 2003 Feb;98(2):428-36. doi: 10.1097/00000542-200302000-00024. PMID 12552203
- [Background] Wunsch H, Kahn JM, Kramer AA, Wagener G, Li G, Sladen RN, Rubenfeld GD. Dexmedetomidine in the care of critically ill patients from 2001 to 2007: an observational cohort study. Anesthesiology. 2010 Aug;113(2):386-94. doi: 10.1097/ALN.0b013e3181e74116. PMID 20613466
- [Background] Pandharipande PP, Pun BT, Herr DL, Maze M, Girard TD, Miller RR, Shintani AK, Thompson JL, Jackson JC, Deppen SA, Stiles RA, Dittus RS, Bernard GR, Ely EW. Effect of sedation with dexmedetomidine vs lorazepam on acute brain dysfunction in mechanically ventilated patients: the MENDS randomized controlled trial. JAMA. 2007 Dec 12;298(22):2644-53. doi: 10.1001/jama.298.22.2644. PMID 18073360
- [Background] Xia ZQ, Chen SQ, Yao X, Xie CB, Wen SH, Liu KX. Clinical benefits of dexmedetomidine versus propofol in adult intensive care unit patients: a meta-analysis of randomized clinical trials. J Surg Res. 2013 Dec;185(2):833-43. doi: 10.1016/j.jss.2013.06.062. Epub 2013 Jul 24. PMID 23910886
- [Background] Alexopoulou C, Kondili E, Diamantaki E, Psarologakis C, Kokkini S, Bolaki M, Georgopoulos D. Effects of dexmedetomidine on sleep quality in critically ill patients: a pilot study. Anesthesiology. 2014 Oct;121(4):801-7. doi: 10.1097/ALN.0000000000000361. PMID 24988068
- [Background] Hughes CG, Girard TD, Pandharipande PP. Daily sedation interruption versus targeted light sedation strategies in ICU patients. Crit Care Med. 2013 Sep;41(9 Suppl 1):S39-45. doi: 10.1097/CCM.0b013e3182a168c5. PMID 23989094
- [Background] Treggiari MM, Romand JA, Yanez ND, Deem SA, Goldberg J, Hudson L, Heidegger CP, Weiss NS. Randomized trial of light versus deep sedation on mental health after critical illness. Crit Care Med. 2009 Sep;37(9):2527-34. doi: 10.1097/CCM.0b013e3181a5689f. PMID 19602975
- [Background] Balzer F, Weiss B, Kumpf O, Treskatsch S, Spies C, Wernecke KD, Krannich A, Kastrup M. Early deep sedation is associated with decreased in-hospital and two-year follow-up survival. Crit Care. 2015 Apr 28;19(1):197. doi: 10.1186/s13054-015-0929-2. PMID 25928417
- [Background] Porhomayon J, Joude P, Adlparvar G, El-Solh AA, Nader ND. The Impact of High Versus Low Sedation Dosing Strategy on Cognitive Dysfunction in Survivors of Intensive Care Units: A Systematic Review and Meta-Analysis. J Cardiovasc Thorac Res. 2015;7(2):43-8. doi: 10.15171/jcvtr.2015.10. PMID 26191390
- [Background] Toft P, Olsen HT, Jorgensen HK, Strom T, Nibro HL, Oxlund J, Wian KA, Ytrebo LM, Kroken BA, Chew M. Non-sedation versus sedation with a daily wake-up trial in critically ill patients receiving mechanical ventilation (NONSEDA Trial): study protocol for a randomised controlled trial. Trials. 2014 Dec 20;15:499. doi: 10.1186/1745-6215-15-499. PMID 25528350
- [Background] Nedergaard HK, Jensen HI, Lauridsen JT, Sjogaard G, Toft P. Non-sedation versus sedation with a daily wake-up trial in critically ill patients receiving mechanical ventilation--effects on physical function: study protocol for a randomized controlled trial: a substudy of the NONSEDA trial. Trials. 2015 Jul 23;16:310. doi: 10.1186/s13063-015-0856-1. PMID 26201718
- [Background] Nedergaard HK, Jensen HI, Stylsvig M, Lauridsen JT, Toft P. Non-sedation versus sedation with a daily wake-up trial in critically ill patients recieving mechanical ventilation - effects on long-term cognitive function: Study protocol for a randomized controlled trial, a substudy of the NONSEDA trial. Trials. 2016 Jun 1;17(1):269. doi: 10.1186/s13063-016-1390-5. PMID 27250658
- [Background] Wu XH, Cui F, Zhang C, Meng ZT, Wang DX, Ma J, Wang GF, Zhu SN, Ma D. Low-dose Dexmedetomidine Improves Sleep Quality Pattern in Elderly Patients after Noncardiac Surgery in the Intensive Care Unit: A Pilot Randomized Controlled Trial. Anesthesiology. 2016 Nov;125(5):979-991. doi: 10.1097/ALN.0000000000001325. PMID 27571256
- [Background] Su X, Meng ZT, Wu XH, Cui F, Li HL, Wang DX, Zhu X, Zhu SN, Maze M, Ma D. Dexmedetomidine for prevention of delirium in elderly patients after non-cardiac surgery: a randomised, double-blind, placebo-controlled trial. Lancet. 2016 Oct 15;388(10054):1893-1902. doi: 10.1016/S0140-6736(16)30580-3. Epub 2016 Aug 16. PMID 27542303
- [Background] International Conference on Harmonisation of technical requirements for registration of pharmaceuticals for human use.. ICH harmonized tripartite guideline: Guideline for Good Clinical Practice. J Postgrad Med. 2001 Jan-Mar;47(1):45-50. No abstract available. PMID 11590294
- [Derived] Sun YM, Zhu SN, Zhang C, Li SL, Wang DX. Effect of low-dose dexmedetomidine on sleep quality in postoperative patients with mechanical ventilation in the intensive care unit: A pilot randomized trial. Front Med (Lausanne). 2022 Aug 31;9:931084. doi: 10.3389/fmed.2022.931084. eCollection 2022. PMID 36117973